CLINICAL TRIAL: NCT00281307
Title: DBPCR Clinical Trial for Treatment of Rhinitis With Intranasal Vitamin E
Brief Title: Treatment of Rhinitis With Intranasal Vitamin E
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to a substantial response to placebo an interim analysis indicated the need for a larger than expected study population to achieve the level of significance
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB 21786
Record Dates: First submitted 2006-01-23; First posted 2006-01-24 (Estimated); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Rhinitis
Keywords: Rhinitis; Vitamin E; Intranasal
MeSH Terms: conditions — Rhinitis

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: RRR-alpha-tocopherol 1,000 IU/mL — Intranasal application three times daily vs. placebo (inert excipient)

SUMMARY:
Many beneficial effects of vitamin E have been described, but vitamin E supplementation by mouth has not been effective in the treatment of nasal symptoms and allergic rhinitis. The investigators will evaluate the effect of vitamin E directly applied to the lining of the nose in individuals with moderate to severe rhinitis by symptom questionnaires.

DETAILED DESCRIPTION:
Vitamin E has health promoting properties that are attributed to its anti-oxidant action and its ability to stabilize cell membrane and promote restoration of the skin barrier function. The beneficial effects of the topical vitamin E applied to the skin have been firmly established and many skin care products now contain vitamin E, whereas the purported benefits cannot be achieved by oral intake of vitamin E. Recently oral vitamin E was shown to be ineffective in the management of allergic rhinitis, which reminisces the clinical experience in dermatology. The failure of oral vitamin E could result from the relatively low local concentration that are not sufficient to scavenge the reactive oxygen species generated in the inflammatory process and restore the consequent epithelial damage to the nasal mucosa in rhinitis.The effect of topical vitamin E applied intranasally to the mucosa has never been studied. It stands to reason that higher local concentrations can be achieved by topical application of vitamin E directly to the nasal mucosa, which may confer the same positive effects observed with its direct application to the skin. We will perform a single center, prospective, randomized, double-blind, placebo-controlled, clinical trial to investigate the role of topical alpha-tocopherol in oil applied to the nasal mucosa 3 times per day with a q-tip on the subjective symptoms of rhinitis over the course of a 4-week period.

ELIGIBILITY:
Inclusion Criteria:

* Clinical symptoms of rhinitis and symptom severity score of 25 or higher on the self-administered Rhinosinusitis Questionnaire (range of 0, i.e. absence of any symptom, to 50, which indicates the most severe symptom in each category)

Exclusion Criteria:

* Inability to give informed consent, comprehend questions or instructions and complete questionnaires
* Recent change (within 2 weeks) in the medications that may affect nasal or sinus symptoms (intranasal or systemic glucocorticosteroids, mast cell stabilizer, antihistamines, decongestants, leukotriene antagonist, antibiotics, preparations containing thyroid or sex hormones, alpha-blocking agents)
* Intranasal use of oil- or gel-based products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2005-12-07 (Actual); Primary Completion 2007-09-01 (Actual); Study Completion 2007-09-01 (Actual)

PRIMARY OUTCOMES:
Reduction in the Rhinitis/Sinusitis Treatment Outcome Questionnaire (ROQa) composite score at the end of the 4th week | 4 weeks

SECONDARY OUTCOMES:
Reduction of severity score for each individual symptom | 4 weeks
Reduction of severity score for the composite symptom score at weekly intervals during the 4-week study period | 4 weeks
Reduction of severity score for the Sinonasal Outcome Test (SNOT-16) at the end of the study | 4 weeks
Reduction of severity score for the Mini-RQLQ (Mini Rhinoconjunctivitis Quality of Life Questionnaire) at the end of the study | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Soheil Chegini, MD, Principal Investigator — Penn State University
Locations (1):
- Cathy Mende, CRNP, Hershey, Pennsylvania, United States

REFERENCES:
- See also: The Human Subjects Protection Office (HSPO) — http://www.hmc.psu.edu/irb